CLINICAL TRIAL: NCT02966054
Title: Self-monitoring and Reminder Texts to Increase Physical Activity After Cancer: a Pilot Randomized Controlled Trial
Acronym: Smart Pace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Erin Van Blarigan, Assistant Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-14452
Record Dates: First submitted 2016-11-09; First posted 2016-11-17 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Colon Cancer; Rectum Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients will be provided with a booklet from the UCSF Dept. of Physical Therapy and Rehabilitation Science: "Moving Through Cancer: A Guide to Exercise for Cancer Survivors". The intervention group will be given a Fitbit® Flex to wear throughout the study and will receive daily text messages to support increased physical activity.
  Interventions: Behavioral: Digital Health Physical Activity Intervention Group
- Control (No Intervention): Patients in the control arm will be provided with a booklet at baseline from the UCSF Dept. of Physical Therapy and Rehabilitation Science: "Moving Through Cancer: A Guide to Exercise for Cancer Survivors".

INTERVENTIONS:
Behavioral: Digital Health Physical Activity Intervention Group — Print materials on exercise after cancer, Fitbit Flex for 12 weeks, and daily Text Messages for 12 weeks
  Arms: Intervention

SUMMARY:
Epidemiologic data consistently indicate that colorectal cancer survivors can improve their quality-of-life and prognosis by engaging in physical activity. This study aims to build on this epidemiologic work and translate the findings to inform and change patient behavior. The specific aims are to: (1) Develop a mobile technology physical activity intervention among colorectal cancer patients who have completed therapy. (2) Conduct a 3-month pilot randomized controlled trial utilizing mobile technology to increase physical activity among 40 men and women who have completed standard cytotoxic chemotherapy for primary stage I-III colorectal cancer at the UCSF Helen Diller Family Comprehensive Cancer Center. Participants in the intervention arm will receive a Fitbit® for self-monitoring, interactive text messages, and educational print materials; participants in the control arm will receive educational print materials at baseline and will be given a Fitbit® after completion of the 3-mo. follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* stage I-III colon or rectal adenocarcinoma
* completed standard cytotoxic chemotherapy if medically indicated
* be considered disease-free at baseline
* be able to speak and read English
* have no contra-indication to moderate to vigorous aerobic exercise
* be able to walk unassisted
* be inactive at baseline (<150 min/week of moderate physical activity)
* have access to a mobile phone
* be able to navigate websites, fill out forms on the web, communicate by email, and have regular access to the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-08; Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Physical activity | 12-weeks
  Change in total physical activity assessed via ActiGraph GT3X+ accelerometers

SECONDARY OUTCOMES:
Fitbit wear time (# days with data / # days of observation) | 12-weeks
Response to text messages (# of messages responded to / # of messages that asked for a response) | 12-weeks
Quality-of-life (SF--36) | 12-weeks
Colorectal cancer-specific quality-of-life (FACT-C) | 12-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Erin Van Blarigan, ScD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Chan H, Van Loon K, Kenfield SA, Chan JM, Mitchell E, Zhang L, Paciorek A, Joseph G, Laffan A, Atreya C, Fukuoka Y, Miaskowski C, Meyerhardt JA, Venook AP, Van Blarigan EL. Quality of life of colorectal cancer survivors participating in a pilot randomized controlled trial of physical activity trackers and daily text messages. Support Care Cancer. 2022 May;30(5):4557-4564. doi: 10.1007/s00520-022-06870-5. Epub 2022 Feb 4. PMID 35119520
- [Derived] Van Blarigan EL, Chan H, Van Loon K, Kenfield SA, Chan JM, Mitchell E, Zhang L, Paciorek A, Joseph G, Laffan A, Atreya CE, Fukuoka Y, Miaskowski C, Meyerhardt JA, Venook AP. Self-monitoring and reminder text messages to increase physical activity in colorectal cancer survivors (Smart Pace): a pilot randomized controlled trial. BMC Cancer. 2019 Mar 11;19(1):218. doi: 10.1186/s12885-019-5427-5. PMID 30866859